CLINICAL TRIAL: NCT01943214
Title: Prospective Cohort Study of the Body Constitution Among Type II Diabetes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Other Study IDs: CE13177
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Body constitution
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Type II DM body constitution: Type II diabetes mellitus, body constitution

SUMMARY:
By analyzing the relationship between the body constitution and the progression of Type II diabetes mellitus, its morbidities, mortality and the impact of the life quality, we try to provide an useful tool, body constitution, to stratify the patients accordingly for individualized health care.

DETAILED DESCRIPTION:
The study participants are recruited from the Diabetes Shared Care Network of the Taichung Veterans General Hospital (Taichung, Taiwan)

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed as Type II diabetes mellitus by Endocrinology specialist.
* aged from 20 to 75 years old.
* clear conscious, willing to join the program.

Exclusion Criteria:

* Severe mental illness, which lead to unable to fulfill the questionaire
* Major surgical intervention,medical events (such as acute myocardial infarction, cerebral vascular accident...et al.,), chemotherapy or radiation therapy within past one month , which made body constitution measurement unavailable.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 type II diabetes mellitus patients recruited from the Endocrinology & Metabolism out patient clinic of Taichung Veterans General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Body constitution of type II diabetes mellitus patients | Two years follow up after being recruited

SECONDARY OUTCOMES:
All cause mortality of type II diabetes mellitus patients | Two years follow up after being recruited
Life quality of diabetes mellitus patients | Two years follow up after being recruited
Diabetic retinopathy of type II diabetes mellitus patients | Two years follow up after being recruited
Diabetic nephropathy of type II diabetes mellitus patients | Two years follow up after being recruited
Diabetic neuropathy of type II diabetes mellitus patients | Two years follow up after being recruited

CONTACTS AND LOCATIONS:
Overall Officials: Chia I Tsai, doctor, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan